CLINICAL TRIAL: NCT05254678
Title: Exercise Rehabilitation Via a Mobile Application for Individuals With Breast Cancer Undergoing Chemotherapy (EMPOWER): A Randomized Controlled Feasibility Trial
Brief Title: Exercise Rehabilitation Via a Mobile Application for Individuals With Breast Cancer Undergoing Chemotherapy
Acronym: Empower
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-21-0429
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Upper Extremity Dysfunction
Keywords: exercise; physical therapy; eHealth
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled feasibility trial
Who Masked: Outcomes Assessor
Masking Description: Independent assessors will be used for collection of objective outcomes. The independent assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard exercise program (Active Comparator): Participants in this group will take part the general exercise program delivered through the Active Living module of the HEAL-ME application. The program comprises (1) supervised group exercise sessions (connection via zoom platform embedded in HEAL-ME), (2) independent exercise workouts within the application, and (3) exercise specific education within the Education Module of the HEAL-ME application.
  Interventions: Behavioral: general exercise
- Integrated physiotherapy and exercise (Experimental): Participants in this group will take part in an integrated physiotherapy and exercise intervention delivered through the Active Living module of the HEAL-ME application. The program comprises (1) supervised group physiotherapeutic exercise sessions (connection via zoom platform embedded in HEAL-ME), (2) independent physiotherapeutic exercise workouts, and (3) breast cancer specific physiotherapy education delivered through weekly modules.
  Interventions: Behavioral: general exercise

INTERVENTIONS:
Behavioral: general exercise — A 10-week integrated physiotherapy and general exercise intervention compared to a general exercise intervention alone.
  Other Names: physiotherapy

SUMMARY:
The primary purpose of this study is to determine the feasibility of our proposed intervention approach involving (1) an integrated physiotherapy and exercise intervention for individuals with breast cancer who are undergoing chemotherapy and (2) delivery of programming via an electronic health (eHealth) application. The secondary objective is to determine the efficacy of the program on upper extremity outcomes, general physical fitness, cancer treatment-related symptoms and quality of life.

DETAILED DESCRIPTION:
EMPOWER is a multi-methods feasibility randomized controlled trial. The study will recruit a minimum of 30 individuals with breast cancer who are undergoing adjuvant chemotherapy following surgery for breast cancer. The study will be conducted in two phases:

Phase I: Randomized Controlled Feasibility Trial The aim of this phase is to determine the feasibility and preliminary efficacy of a 10-week integrated physiotherapy and exercise intervention compared to an exercise intervention alone.

Phase II: Qualitative Study The aim of this phase is to evaluate the acceptability of the Healthy Eating, Active Living and Mindful Energy (HEAL-ME) Research App design, program delivery, program components and perceived effectiveness of the intervention at the level of the participant.

PHASE I: Randomized Controlled Feasibility Trial A randomized controlled trial design will be used to randomize individuals with breast cancer to one of two groups: 1) Comparison group: general exercise intervention + education; and 2) Experimental group: integrated physiotherapy and general exercise intervention + education. The study will be carried out over a 10-week period. The outcome measures will be assessed at baseline and at 10 weeks.

Randomization: An independent researcher will generate the randomization sequence using a computer-generated randomization module within the Trial's REDCap database. Randomization will occur following baseline testing.

Interventions:

Group 1 (Comparator): Hybrid In-Persona and HEAL-ME delivered General Exercise:

Participants in this group will take part the general exercise program delivered in-person and through the Active Living module of the HEAL-ME application. The program comprises (1) supervised group exercise sessions in-person or virtually (2) independent exercise workouts within the application, and (3) exercise specific education within the Education Module of the HEAL-ME application. Exercise regimen: The exercise regimen follows the general principles of overload, progression, and specificity. The exercise program consists of full body exercise (e.g., comprising aerobic, resistance training, core stability, balance and flexibility training) a minimum of 2 times per week (one group virtual session and one independent self-directed session). Education: educational materials in written (PDF format) will be included in the Education module: resources section of the HEAL-ME application. Topics include the exercise expectations, behavior change strategies, home exercise equipment and how to exercise safely.

Group 2 (Experimental): Hybrid in-person and HEAL-ME Integrated Physiotherapy and exercise:

Participants in this group will take part in an integrated physiotherapy and exercise intervention delivered in-person and through the Active Living module of the HEAL-ME application. The program comprises (1) supervised group physiotherapeutic exercise sessions in-person or virtually, (2) independent physiotherapeutic exercise workouts, and (3) breast cancer specific physiotherapy education delivered through weekly modules. Integrated physiotherapy and exercise regimen: The integrated physiotherapy and exercise regimen will follow the exercise regimen as described in Group 1. For this group, breast cancer specific shoulder range of motion and stretching exercises will be incorporated into the warm-up and cool-down components of both group and individual exercise sessions. Education: educational videos will be available on the application and include topics such as cancer-related fatigue, risk reduction for lymphedema and pelvic health after breast cancer.

Educational materials in written (PDF format) will be included in the Education module: resources section of the HEAL-ME application. Topics include the benefits of exercise during chemotherapy for breast cancer, exercise behavior change strategies, and how to exercise safely.

Blinding An independent assessor, who is blinded to the group assignment will carry out all the measurements. Training of the assessor will be conducted on the measurement procedures related to the upper body and fitness outcome measurement protocols prior to study initiation.

PHASE II: Assessment of HEAL-ME App Design, Acceptability, and Program Components The app design, acceptability, and program components will be assessed following completion of the study through focus groups and semi-structured interviews to explore the experiences of individuals randomized to the HEAL-ME experimental group. The purpose of this phase is to assess different aspects of HEAL-ME related to the program delivery, different components contents, and time commitment. The results of this phase will inform further development of the HEAL- ME breast cancer module.

Phase II Data Collection Focus Groups: E-intervention group participants will be invited to participate in a focus group or semi-structured interview session that aim to capture participant perspectives and experiences, as well as any facilitators or barriers to use of the HEAL-ME application.

Qualitative Data Analysis The focus groups discussions will be audio recorded and transcribed. Two researchers will read and then reread the transcripts for accuracy against the audio recordings. The investigators will conduct an inductive content analysis to capture the participants' views about the program's acceptability and usability and ways to refine it. The inductive approach will enable a descriptive evaluation of the program from the participant's view. Two researchers will independently analyze the content of the focus group transcripts to identify evidence related to research objectives. Using the thematic analytic approach, the investigators will follow different processes described by Braun and Clarke. The data will be analyzed line by line by the researchers independently to identify patterns and key themes with example quotes from the data. Codes for similar meanings and highlighted terms will be developed, examined, and refined if necessary to identify the most expressive codes related to the research objectives. The process will be repeated a few times until concrete themes emerge and no further themes are identified. The generated themes will be reviewed and verified by a third researcher in order to increase the validity of the findings. Any coding discrepancies will be discussed and reconciled. Conceptual themes will be inductively originated from analysis through generating initial codes, followed by sub-themes, and finally, an overarching theme.

ELIGIBILITY:
Inclusion Criteria:

* adult females with a diagnosis of breast cancer (Stage Ic-III);
* be able to participate in mild levels of activity at minimum;
* have completed cancer surgery involving a mastectomy or breast conserving surgery involving either an axillary lymph node dissection or sentinel lymph node biopsy;
* having completed or undergoing adjuvant chemotherapy +/- biological therapy treatment (eligible from 4 weeks to one year post-surgery at baseline);
* speak and understand English.

Exclusion Criteria:

* unable to commit to the 10-week virtual program including testing sessions at the Cancer Rehabilitation clinic in the Corbett Hall at the University of Alberta;
* do not have regular access to the internet and a smart device or computer in the home.
* are scheduled to undergo neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Completion rate | 10 weeks
  Defined as >70% participants completing at least 70% of exercise sessions and the post-study assessment

SECONDARY OUTCOMES:
Recruitment rate | one year
  Percentage of participants eligible who consent to participate in the study
Attendance rate | 10 weeks
  Percentage of completed exercise and education modules
Program Satisfaction | 10 weeks
  Program Satisfaction Questionnaire
Symptoms | 10 weeks
  Edmonton Symptom Assessment System
Health-related Quality of Life | 10 weeks
  Functional Assessment of Cancer Therapy -breast (FACT-B+4)
Fatigue | 10 weeks
  Functional Assessment of Cancer Therapy - fatigue subscale (FACIT-F)
Physical Activity | 10 weeks
  Godin Leisure Time Exercise Questionnaire
Cost-effectiveness | 10 weeks
  EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Walking endurance | 10 weeks
  Six-minute walk test
Lower body strength | 10 weeks
  Thirty second sit-to-stand
Flexibility Shoulder Flexion | 10 weeks
  Active Shoulder Range of Motion: flexion
Flexibility Shoulder Abduction | 10 weeks
  Active Shoulder Range of Motion: abduction
Flexibility Shoulder External Rotation | 10 weeks
  Active Shoulder Range of Motion: external rotation
Flexibility Shoulder Internal Rotation | 10 weeks
  Active Shoulder Range of Motion: internal rotation
Flexibility Shoulder Horizontal Abduction | 10 weeks
  Active Shoulder Range of Motion: horizontal abduction
Flexibility lower body | 10 weeks
  Sit-and-reach
Balance | 10 weeks
  One-leg Stance Test
Arm volume | 10 weeks
  Perometry for the measurement of lymphedema
Body weight | 10 weeks
  Measurement of weight in kgs
Body height | 10 weeks
  Measurement of height in cms

OTHER OUTCOMES:
Grip strength (optional) | 10 weeks
  Dynamometry
Core muscular endurance (optional) | 10 weeks
  Plank endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
On completion of the trial, data will be available through the University of Alberta's Dataserve
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When study findings have been published
Access Criteria: The data on repository will be available on request to the principal investigator.